CLINICAL TRIAL: NCT02400736
Title: Efficacy of Supported Employment Within the OIF/OEF Patient Aligned Care Team
Brief Title: Supported Employment in Patient Aligned Care Teams
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1489-I
Record Dates: First submitted 2015-03-10; First posted 2015-03-27 (Estimated); Results first posted 2021-03-30 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Mental Disorder; Substance Use Disorders; Posttraumatic Stress Disorder; Major Depressive Disorder; Anxiety Disorder
Keywords: Veterans; Patient Aligned Care Team; Primary Care; Mental Disorders; Substance Use Disorders; Posttraumatic Stress disorder; Major Depression; Individual Placement and Support; Supported Employment; Vocational Rehabilitation; Transitional Work; Anxiety Disorders
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders; Stress Disorders, Post-Traumatic; Depressive Disorder, Major; Anxiety Disorders | interventions — Palliative Care; Employment, Supported; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individual Placement and Support (IPS) (Experimental): Individual Placement and Support (IPS) is supported employment and involves the following domains: 1) competitive employment: IPS assists participants to enter into competitive jobs; 2) eligibility based on client choice, i.e. "zero exclusion"; 3) integration of IPS and treatment team, i.e. the PACT; 4) patient-centered job match for competitive employment; 5) personalized benefits counseling: IPS specialists help Veterans obtain information about their VA, Social Security, Medicaid, and other government entitlements; 6) rapid job search: IPS specialists use a rapid job search, rather than providing lengthy pre-employment assessment, training, counseling; 7) job development: IPS specialists build an employer network based on Veterans' interests; 8) time-unlimited and individualized support: follow-along IPS supports are individualized and continue for as long as needed during the 12-month study.
  Interventions: Behavioral: Individual Placement and Support (IPS)
- Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR) (Active Comparator): Treatment as Usual Vocational Rehabilitation includes pre-vocational counseling, Community Based Supported Employment, or most commonly Transitional Work assignments (TW) which involves 1) time-limited set-aside work experiences: short-term transitional work experiences in a brokered or set-aside work setting; 2) no strict entrance criteria other than general medical clearance; 3) limited integration of TW and clinical Services; 4) not patient-centered: TW jobs are pre-arranged, set-aside jobs are less likely to have a meaningful relationship to the Veterans' preferences; 5) personalized benefits counseling; 6) limited job search: TW specialists provide variable and limited guidance for competitive job search; 7) no job development: TW specialists do not engage in community based job development; 8) time limited: The TW specialist does not provide long-term follow-up after the first job is obtained.
  Interventions: Other: Treatment as Usual Vocational Rehabilitation/Transitional Work (TUA-VR)

INTERVENTIONS:
Behavioral: Individual Placement and Support (IPS) — Individual Placement and Support (IPS) is the evidenced based model of supported employment.
  Other Names: Supported Employment
  Arms: Individual Placement and Support (IPS)
Other: Treatment as Usual Vocational Rehabilitation/Transitional Work (TUA-VR) — Vocational Rehabilitation Treatment as Usual includes pre-vocational counseling, Community Based Supported Employment, or most commonly Transitional Work assignments (TW).
  Other Names: Treatment as Usual; Transitional Work
  Arms: Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR)

SUMMARY:
In response to the Rehabilitation Research and Development (RR&D) Deployment Health Research, this study addresses the delivery of an evidenced-based vocational rehabilitation, specifically Individual Placement and Support (IPS), for Veterans who are facing unemployment and mental illness as they try to recovery and re-establish civilian life. This study provides the requisite evidence needed to guide the Veterans Health Administration (VHA) as to whether to expand the target population for IPS to Veterans with any mental disorder, delivered directly within the primary care setting (i.e. Patient Aligned Care Team; PACT). Such modifications in VHA practice could substantially improve Veteran vocational rehabilitation access and outcomes, moving a significantly greater number of disabled Veterans back to full and productive lives in the community.

DETAILED DESCRIPTION:
Background: Veterans returning from Iraq and Afghanistan wars often confront unemployment as they reintegrate into civilian life. Over the past two decades, studies of Individual Placement and Support (IPS) supported employment have yielded remarkably robust and consistent vocational rehabilitation outcomes. However, IPS has predominantly only been studied in mental health settings and in the seriously mentally ill populations. Access to a mental health setting for recently deployed Veterans is often delayed by months or years, and thus, result in substantial delay of referrals to vocational rehabilitation programs which leave many Veterans vulnerable to continued unemployment and a deteriorating trajectory.

Methods: This single site, prospective, randomized, controlled study evaluated the efficacy of IPS when delivered within primary care Patient Aligned Care Teams (PACT). Participants were U.S. military Veterans who served in the Operation Enduring Freedom, Operation Iraqi Freedom, and Operation New Dawn (OEF/OIF/OND) and/or any other Southwest Asia operations (i.e. since 1990) who were receiving care in a primary care PACT, currently unemployed and diagnosed with any mental disorder other than a serious mental illness. Eligible participants were randomized 1:1 to either IPS or VHA treatment as usual vocational rehabilitation (TAU-VR) which included prevocational counseling, community based supported employment, or most commonly Transitional Work assignment. Compared to TAU-VR (control condition), IPS delivered within a PACT was hypothesized to result in a higher rate of steady workers, as defined by working >/=50% of the weeks in the 12-month follow-up period in a competitive job (primary outcome), more weeks worked in a competitive job, and more income earned.

Significance: In an innovative approach, this study breaks from the diagnostic categorical approach and the mental health treatment setting and evaluates the efficacy of IPS when delivered in a primary care setting, specifically a PACT that serves Veterans who have returned from the Iraq, Afghanistan, and other Southwest Asia conflicts. Making a substantial paradigm shift, this study integrates IPS within a PACT for the first time ever. The research is directly linked to the RR&D priority areas of improving vocational outcomes and promoting recovery in Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Age 19* (<19 years of age is the state of Alabama defined minor)
* Receiving primary care treatment in the Tuscaloosa VA Medical Center (TVAMC) PACT, called the Transition Center (i.e. served during the OEF/OIF/OND/other Southwest Asia conflicts) or other Primary Care PACT providing care for OEF/OIF/OND/other Southwest Asia Veteran
* Otherwise eligible for TVAMC vocational rehabilitation services, in the event that the Veteran is randomized to TW
* diagnosis that is disabling or potentially disabling (i.e. depressive, bipolar II, anxiety, obsessive-compulsive, trauma- and stressor-related, dissociative, impulse- control, and substance related/addictive (other than caffeine and nicotine) disorder classifications), other than those listed as exclusionary, within past 90 days according to Diagnostic and Statistical Manual 5th edition.
* Currently unemployed, defined as not working in a competitive job for a wage or under-employed, defined as (defined as: working less than 20 hours per week in a job that is low wage and is not in keeping with the Veteran's ability, aptitude, or skills)
* Expression of interest in competitive employment
* Willing and able to give informed consent.

Note: Veterans with history of mild traumatic brain injury (TBI) may be included in the study.

Exclusion Criteria:

* Current diagnosis of (i) schizophrenia, (ii) schizoaffective, (iii) bipolar I disorder, or major depression with psychotic features, since these Veterans may receive IPS in mental health
* Diagnosis of dementia (evidenced in the medical record)
* Clinically significant unstable or severe medical condition, or terminal illness, that would contraindicate study participation or expose them to an undue risk of a significant adverse event
* Unlikely that participant can complete the study, e.g. expected deployment, incarceration, long-term hospitalization, or relocation from the vicinity of the TVAMC during the study period
* Active suicidal or homicidal ideation making it unsafe for Veteran to be included in study
* Current participation in another interventional trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori L Davis, MD, Principal Investigator — Tuscaloosa VA Medical Center, Tuscaloosa, AL
Locations (1):
- Tuscaloosa VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared.

REFERENCES:
- [Background] Davis LL, Blansett CM, Mumba MN, MacVicar D, Toscano R, Pilkinton P, Gay W, Bartolucci A. The methods and baseline characteristics of a VA randomized controlled study evaluating supported employment provided in primary care patient aligned care teams. BMC Med Res Methodol. 2020 Feb 17;20(1):33. doi: 10.1186/s12874-020-0919-1. PMID 32066380
- [Derived] Davis LL, Mumba MN, Toscano R, Pilkinton P, Blansett CM, McCall K, MacVicar D, Bartolucci A. A Randomized Controlled Trial Evaluating the Effectiveness of Supported Employment Integrated in Primary Care. Psychiatr Serv. 2022 Jun;73(6):620-627. doi: 10.1176/appi.ps.202000926. Epub 2021 Sep 15. PMID 34521208
- See also: Methods and Baseline paper — http://doi.org/10.1186/s12874-020-0919-1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 502 veterans were considered for this study, 140 were consented, 19 were not eligible, 2 were randomized in error, and 119 were randomized and included in the analyses. Of the 119 randomized participants, 100 (84%) participants completed the study.
Groups:
- Individual Placement and Support (IPS): .Individual Placement and Support (IPS) is supported employment and involves the following domains: 1) competitive Employment: IPS assists participants to enter into competitive jobs; 2) eligibility based on client choice, i.e. "zero exclusion"; 3) integration of IPS and treatment team, i.e. the Patient Aligned Care Team (PACT); 4) patient-centered job match for competitive employment; 5) personalized benefits counseling: IPS specialists help Veterans obtain information about their VA, Social Security, Medicaid, and other government entitlements; 6) rapid job search: IPS specialists use a rapid job search, rather than providing lengthy pre-employment assessment, training, counseling; 7) job development: IPS specialists build an employer network based on Veterans' interests; 8) time-unlimited and individualized support: follow-along IPS supports are individualized and continue for as long as needed during the 12-month study.
- Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR): Treatment as Usual Vocational Rehabilitation could include pre-vocational counseling, Community Based Supported Employment, and most commonly Transitional Work assignments (TW) which involves 1) time-limited set-aside work experiences: short-term transitional work experiences in a brokered or set-aside work setting; 2) no strict entrance criteria other than general medical clearance; 3) limited integration of TW and clinical Services; 4) not patient-centered: TW jobs are pre-arranged, set-aside jobs are less likely to have a meaningful relationship to the Veterans' preferences; 5) personalized benefits counseling; 6) limited job search: TW specialists provide variable and limited guidance for competitive job search; 7) no job development: TW specialists do not engage in community based job development; 8) time limited: The TW specialist does not provide long-term follow-up after the first job is obtained.
Period: Overall Study
Arm/Group | Individual Placement and Support (IPS) | Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR)
Started | 58 | 61
Completed | 47 | 53
Not Completed | 11 | 8
Not completed — Lost to Follow-up | 6 | 6
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Moved from the area | 3 | 1

BASELINE CHARACTERISTICS:
Population: 140 Veterans were consented and 119 Veterans were randomized and included in the analysis. Two were randomized randomized in error and were not included in the analysis. For the 19 not randomized, 4 had no qualifying DSM-5 diagnosis, 5 changed their mind, 3 were unlikely to complete, 2 were employed; 3 were not eligible for vocational rehabilitation services; 1 declined competitive employment; 1 was enrolled in another interventional study.
Groups:
- Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR): Treatment as Usual Vocational Rehabilitation could include pre-vocational counseling, Community Based Supported Employment, and most commonly Transitional Work assignments (TW) which involves 1) time-limited set-aside work experiences: short-term transitional work experiences in a brokered or set-aside work setting; 2) no strict entrance criteria other than general medical clearance; 3) limited integration of TW and clinical Services; 4) not patient-centered: TW jobs are pre-arranged, set-aside jobs are less likely to have a meaningful relationship to the Veterans' preferences; 5) personalized benefits counseling; 6) limited job search: TW specialists provide variable and limited guidance for competitive job search; 7) no job development: TW specialists do not engage in community based job development; 8) time limited: TW specialist does not provide long-term follow-up after the first job is obtained.
- Total: Total of all reporting groups
Arm/Group | Individual Placement and Support (IPS) | Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR) | Total
Number analyzed (Participants) | 58 | 61 | 119
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 37.8 (8.4) | 38.6 (8.4) | 38.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 49 | 49 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 57 | 60 | 117
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 42 | 45 | 87
  White | 15 | 16 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Mental Disorder [Count of Participants; unit: Participants] — MINI International Neuropsychiatric Interview Version 7 (MINI) to assess concurrent mental disorders for Diagnostic and Statistical Manual Fifth Edition (DSM-5). A participant could have more than one diagnosis, i.e. number of disorders exceeds number of participants
  Participants
    Major depression, past | 49 | 48 | 97
    Major depression, current | 43 | 41 | 84
    Agoraphobia | 7 | 13 | 20
    Panic Disorder (lifetime) | 24 | 27 | 51
    Post-traumatic stress disorder | 46 | 44 | 90
    Alcohol Use Disorder, past year | 29 | 26 | 55
    Substance Used Disorder | 29 | 27 | 56

OUTCOME MEASURES:

1. Primary Outcome: Steady Worker
Description: Participants were categorized as a steady worker if they held a competitive job for 50% or more of the 12-month follow-up (i.e. 26 or more weeks out of 52 weeks).
Time Frame: 12 months
Population: 119 randomized Veterans who were followed in a primary care Patient Aligned Care Team, who had a diagnosis of at least one mental disorder, and were unemployed or under-employed.
Measure: Count of Participants; unit: Participants
Groups:
- Individual Placement and Support (IPS): Individual Placement and Support (IPS) is supported employment and involves the following domains: 1) competitive Employment: IPS assists participants to enter into competitive jobs; 2) eligibility based on client choice, i.e. "zero exclusion"; 3) integration of IPS and treatment team, i.e. the Patient Aligned Care Team; 4) patient-centered job match for competitive employment; 5) personalized benefits counseling: IPS specialists help Veterans obtain information about their VA, Social Security, Medicaid, and other government entitlements; 6) rapid job search: IPS specialists use a rapid job search, rather than providing lengthy pre-employment assessment, training, counseling; 7) job development: IPS specialists build an employer network based on Veterans' interests; 8) time-unlimited and individualized support: follow-along IPS supports are individualized and continue for as long as needed during the 12-month study.
Arm/Group | Individual Placement and Support (IPS) | Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR)
Number analyzed (Participants) | 58 | 61
Participants | 26 | 15
Statistical Analysis 1: Comparison: Individual Placement and Support (IPS) vs Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR); Using SamplePower 3.0 to estimate the statistical power, the target sample size of 120 (60 per group) provided 84% power to detect a 25% or greater absolute difference between groups in the percent of participants achieving 'steady worker' status (e.g., 40% in IPS vs. 15% in control arm), at the .05 level of significance, assuming a 10% attrition; Test type: Superiority — Proportion of steady workers in each group was analyzed using a logistic regression model to calculate an odds ratio and 95% Confidence Interval. Adhering to the principle of intent-to-treat, participants were retained in the arm to which they were randomized for the 12-month follow-up period despite discontinuing the treatment intervention or exiting the study early. Missing data was counted as "not worked."; p = 0.02, Chi-squared — a priori threshold for statistical significance p </=0.05; not adjusted for multiple comparisons; Odds Ratio (OR) = 2.49, 95% CI 2-sided [1.14 to 5.43]

2. Secondary Outcome: Weeks Worked in a Competitive Job
Description: Number of weeks out of 52 week follow-up in which the participant worked at least one hour in a competitive job.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Individual Placement and Support (IPS) | Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR)
Number analyzed (Participants) | 58 | 61
weeks | 38.6 (14.8) | 24.6 (17.2)
Statistical Analysis 1: Comparison: Individual Placement and Support (IPS) vs Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR); Total mean time worked was compared using an analysis of variance (ANOVA); Test type: Superiority — Intent to treat analysis; p = 0.003, t-test, 2 sided — a priori threshold for statistical significance p </=0.05; not adjusted for multiple comparisons

3. Secondary Outcome: Time to First Competitive Job
Description: The number of weeks from randomization until the participant worked in a competitive job.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Individual Placement and Support (IPS) | Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR)
Number analyzed (Participants) | 58 | 61
weeks | 8.7 (8.8) | 17.6 (14.2)
Statistical Analysis 1: Comparison: Individual Placement and Support (IPS) vs Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR); intent to treat analysis; Test type: Superiority; p = 0.005, Mixed Models Analysis — a priori threshold for statistical significance p </=0.05; not adjusted for multiple comparisons

4. Secondary Outcome: Income Earned From Competitive Jobs
Description: For those participants, the income earned from any competitive jobs was added for the 52-week follow-up period.
Time Frame: 12 months
Population: Randomized participants
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | Individual Placement and Support (IPS) | Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR)
Number analyzed (Participants) | 58 | 61
US dollars | 11,106 (12,792) | 6,605 (10,150)
Statistical Analysis 1: Comparison: Individual Placement and Support (IPS) vs Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR); Test type: Superiority — a priori threshold for statistical significance p </=0.05; not adjusted for multiple comparisons; p = 0.033, t-test, 2 sided

5. Secondary Outcome: Symptom Checklist-90-Revised Change From Baseline to Month 12.
Description: Symptom Checklist-90-Revised (SCL-90-R): 90-item self-report survey; assesses nine dimensions. Each item is self-rated for level of discomfort/distress on scale of 0 "not at all" to 4 "extremely" for somatization (range 0 to 48), obsessive-compulsive symptoms (range 0 to 40), interpersonal sensitivity (range 0 to 36), depression (range 0 to 52), anxiety (range 0 to 40), hostility (range 0 to 24), phobic-anxiety (range 0 to 28), paranoid ideation (range 0 to 24), and psychoticism (range 0 to 40). Total score for a dimension is the sum of items and the distress score for each dimension is the sum divided by number of items in that dimension (range = 0 to 4). Global Severity Index is a mean of all items, calculated by dividing the sum of scores by the number of items (range 0 to 4). Higher score indicates greater distress and increase in score over time indicates worse outcome.
Time Frame: Change from baseline to month 12 (value at 12 months minus value at baseline) is shown below. Additionally, all relevant time points used in the calculation timeframe from baseline to 12 months (baseline, months 4, 6, 8, and 12) included in analysis.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individual Placement and Support (IPS) | Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR)
Number analyzed (Participants) | 58 | 61
score on a scale | 0.036 (0.14) | 0.042 (0.15)
Statistical Analysis 1: Comparison: Individual Placement and Support (IPS) vs Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR); Test type: Superiority; p = 0.853, Mixed Models Analysis — a priori threshold for statistical significance p </=0.05; not adjusted for multiple comparisons; Effect of treatment on outcome was analyzed using longitudinal mixed-effects regression model.Group by time interaction tested for treatment effect

6. Secondary Outcome: Income Earned From All Sources
Description: All income earned from competitive, transitional work, and other sources over the 12-month follow-up.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | Individual Placement and Support (IPS) | Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR)
Number analyzed (Participants) | 58 | 61
US dollars | 17,960 (11,310) | 11,168 (9,682)
Statistical Analysis 1: Comparison: Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR); Test type: Superiority — a priori threshold for statistical significance p </=0.05; not adjusted for multiple comparisons; p = 0.004, t-test, 2 sided

7. Secondary Outcome: Rosenberg Self-Esteem Scale Change From Baseline to 12 Months.
Description: Rosenberg Self-Esteem Scale (RSES) is a 10-item self-report Likert-type questionnaire that asks participants to indicate the degree of their agreement or disagreement with statements about their self-esteem and self-depreciation from 0 = "strongly agree" to 3 = "strongly disagree". The items are summed and the scoring ranges from 0 to 30, with higher scores indicating a higher degree of self-esteem; a positive change in score over time indicates improved self esteem. A score less than 15 may indicate low self esteem.
Time Frame: Change from baseline to month 12 (value at 12 months minus value at baseline) is shown below. Additionally, all relevant time points used in the calculation timeframe from baseline to 12 months (baseline, months 4, 6, 8, 12) were included in mixed model.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individual Placement and Support (IPS) | Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR)
Number analyzed (Participants) | 58 | 61
score on a scale | 1.23 (5.16) | 0.31 (6.33)
Statistical Analysis 1: Comparison: Individual Placement and Support (IPS) vs Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR); The effect of treatment on each of secondary outcome measures were analyzed using a longitudinal mixed-effects regression model. The group by time interaction tested for the treatment effect; Test type: Superiority; p = 0.47, Mixed Models Analysis — a priori threshold for statistical significance p </=0.05; not adjusted for multiple comparisons; [statistical method as in outcome 5, analysis 1]

8. Secondary Outcome: Income Earned From Competitive Jobs in Participants Who Held a Competitive Job
Description: Income earned ($) from competitive jobs over 12 months was compared between groups for all randomized participants who held a competitive job at some point.
Time Frame: 12 months
Population: All randomized participants who held a competitive job during the 12-month follow-up
Measure: Mean (Standard Deviation); unit: US dollars
Groups:
- Individual Placement and Support (IPS): .Individual Placement and Support (IPS) is supported employment and involves the following domains: 1) competitive Employment: IPS assists participants to enter into competitive jobs; 2) eligibility based on client choice, i.e. "zero exclusion"; 3) integration of IPS and treatment team, i.e. the Patient Aligned Care Team; 4) patient-centered job match for competitive employment; 5) personalized benefits counseling: IPS specialists help Veterans obtain information about their VA, Social Security, Medicaid, and other government entitlements; 6) rapid job search: IPS specialists use a rapid job search, rather than providing lengthy pre-employment assessment, training, counseling; 7) job development: IPS specialists build an employer network based on Veterans' interests; 8) time-unlimited and individualized support: follow-along IPS supports are individualized and continue for as long as needed during the 12-month study.
Arm/Group | Individual Placement and Support (IPS) | Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR)
Number analyzed (Participants) | 36 | 31
US dollars | 18,945 (10,792) | 13,813 (10,809)
Statistical Analysis 1: Comparison: Individual Placement and Support (IPS) vs Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR); Test type: Superiority; p = 0.062, t-test, 2 sided — a priori threshold for statistical significance p </=0.05; not adjusted for multiple comparisons

9. Other Pre Specified Outcome: Community Reintegration of Service Members
Description: Community Reintegration of Service Members (CRIS) is a self-report instrument used to evaluate the Veteran's reintegration into the community. The correlations between the CRIS and the 36-Item Short Form Health Survey scales of role physical, role emotional, and social functioning were 0.44-0.80 and the CRIS has strong reliability, conceptual integrity, and construct validity. In pilot studies with 126 veterans, working subjects had better CRIS scores then unemployed subjects. Items on the CRIS cover 9 aspects of participation: Learning and Applying Knowledge, General Tasks and Demands, Communication, Mobility, Self-care, Domestic Life, Interpersonal Relationships, Major Life Areas, and Community, Social and Civic Life. Subscale scores for 1) extent of participation, 2) perceived limitations, and 3) satisfaction with participation are calculated. For each of the 3 subscales, the minimum score is 10, the maximum score is 70. Higher scores are indication of better outcomes.
Time Frame: 12 months
Population: All subjects randomized; intent-to-treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Individual Placement and Support (IPS) | Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR)
Number analyzed (Participants) | 58 | 61
units on a scale
  Baseline (Extent of Participation) | 46.8 (8.15) | 48.6 (7.75)
  4-month (Extent of Participation): number analyzed (Participants) | 32 | 45
  4-month (Extent of Participation) | 48.6 (6.32) | 48.5 (7.98)
  8-month (Extent of Participation): number analyzed (Participants) | 32 | 40
  8-month (Extent of Participation) | 48.1 (7.51) | 46.3 (8.55)
  12-month (Extent of Participation): number analyzed (Participants) | 38 | 48
  12-month (Extent of Participation) | 46.1 (8.61) | 47.6 (9.50)
  Baseline (Perceived Limitations) | 47.1 (8.77) | 48.0 (7.34)
  4-month (Perceived Limitations): number analyzed (Participants) | 32 | 45
  4-month (Perceived Limitations) | 49.9 (7.96) | 48.7 (8.81)
  8-month (Perceived Limitations): number analyzed (Participants) | 32 | 40
  8-month (Perceived Limitations) | 47.8 (8.97) | 47.7 (9.01)
  12-month (Perceived Limitations): number analyzed (Participants) | 38 | 48
  12-month (Perceived Limitations) | 46.7 (9.21) | 48.1 (9.82)
  Baseline (Satisfaction with Participation) | 48.6 (9.89) | 50.6 (9.91)
  4-Month (Satisfaction with Participation): number analyzed (Participants) | 32 | 45
  4-Month (Satisfaction with Participation) | 52.6 (8.62) | 51.7 (9.34)
  8-month (Satisfaction with Participation): number analyzed (Participants) | 32 | 40
  8-month (Satisfaction with Participation) | 50.3 (10.11) | 50.2 (10.92)
  12-month (Satisfaction with Participation): number analyzed (Participants) | 38 | 48
  12-month (Satisfaction with Participation) | 47.7 (10.11) | 50.4 (11.45)
Statistical Analysis 1: Comparison: Individual Placement and Support (IPS) vs Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR); Test type: Superiority; p > 0.3, ANOVA — a priori threshold for statistical significance p </= 0.05 or lower. No adjustments were made for multiple comparisons

10. Post Hoc Outcome: Proportion of Weeks Unencumbered by Transitional Work in Which Competitive Job Was Held
Description: The number of weeks in which the participant was engaged in a transitional work assignment in the treatment as usual arm was subtracted from the 52 week follow-up and used as denominator in deriving the proportion of weeks worked in a competitive job. The IPS group did not engage in transitional work, so 52 weeks was the denominator in deriving the proportion of weeks worked in a competitive job.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of 52 weeks
Arm/Group | Individual Placement and Support (IPS) | Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR)
Number analyzed (Participants) | 58 | 61
percentage of 52 weeks | 40 (13.7) | 25 (16.7)
Statistical Analysis 1: Comparison: Individual Placement and Support (IPS) vs Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR); Test type: Superiority; p = 0.001, t-test, 2 sided — a priori threshold for statistical significance p </=0.05; not adjusted for multiple comparisons

11. Post Hoc Outcome: Held a Full-time Competitive Job
Description: Participant held a full-time competitive job during the 12-month follow-up. Full time was defined as working at least 30 hours per week.
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Individual Placement and Support (IPS) | Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR)
Number analyzed (Participants) | 58 | 61
Participants | 25 | 12
Statistical Analysis 1: Comparison: Individual Placement and Support (IPS) vs Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR); Test type: Superiority; p = 0.006, Chi-squared — a priori threshold for statistical significance p </=0.05; not adjusted for multiple comparisons

ADVERSE EVENTS:
Time Frame: 12 months
Description: Participants self-reported adverse events were collected over 12-months and definition did not differ from clinical trials site. Adverse events were monitored without regard to the specific adverse event term.
Arm/Group | Individual Placement and Support (IPS) | Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR)
All-Cause Mortality (participants affected / at risk) | 1/58 | 0/61
Serious Adverse Events (participants affected / at risk) | 6/58 | 4/61
Other Adverse Events (participants affected / at risk) | 17/58 | 22/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individual Placement and Support (IPS) (N=58) | Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR) (N=61)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) — Hospitalized for Seizures
Suicidal Ideation (Psychiatric disorders) | 2 (2) | 1 (1) — Hospitalized for suicidal ideation and depression.
Kidney Stone (Renal and urinary disorders) | 1 (1) | 0 (0) — Hospitalize due to pain from kidney stone
Gun Shot Wound (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Hospitalized for observation.
Peptic Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) — Hospitalized for chest pain but determined cause was acid reflux and peptic ulcer
Death (Cardiac disorders) | 1 (1) | 0 (0) — Death due to myocardial infarction
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Hospitalized for prostate cancer
Chest Pain (Cardiac disorders) | 1 (2) | 0 (0) — hospitalized due to chest pain
Hysterectomy (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Hospitalized for hysterectomy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individual Placement and Support (IPS) (N=58) | Treatment as Usual Vocational Rehabilitation/Transitional Work (TAU-VR) (N=61)
Muscular Skeletal Pain or Problem (Musculoskeletal and connective tissue disorders) | 8 (10) | 9 (11)
Infection (Infections and infestations) | 3 (3) | 6 (7) — Viral an/d bacterial
Mental health (Psychiatric disorders) | 2 (2) | 1 (1) — mental health or substance use
Eye (Eye disorders) | 1 (1) | 1 (1) — Problems pertaining to eye.
Neurological (Nervous system disorders) | 2 (2) | 4 (4) — Headache, spinal disc problem, or Seizure
Cardiovascular (Cardiac disorders) | 1 (1) | 1 (1)
Reproductive system (Reproductive system and breast disorders) | 1 (1) | 1 (1)
GI, including dental (Gastrointestinal disorders) | 1 (1) | 2 (2)
Ear (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Pmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Accidents, insects, dog bites (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Diabetes (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations: single-site, veterans only, under representation of women, and the site only achieved "fair" level of implementation of IPS based on the IPS Fidelity Scale. Transitional work assignments may have weakened employment outcomes in control group; but only half of the control group held a TW assignment. Strengths: randomized approach, credible control group, 12-month follow-up, broad eligibility criteria, and novel setting (i.e. primary care setting).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-02): https://cdn.clinicaltrials.gov/large-docs/36/NCT02400736/Prot_SAP_000.pdf